CLINICAL TRIAL: NCT00389428
Title: Phase 1 Study of CPX-351(Cytarabine:Daunorubicin) Liposome Injection in Patients With Advanced Hematologic Malignancies.
Brief Title: Multicenter Study of CPX-351(Cytarabine:Daunorubicin) Liposome Injection in Patients With Advanced Hematologic Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0305-101
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic malignancies; Malignancies, hematologic; Hematopoietic malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — CPX-351; Liposomes

INTERVENTIONS:
Drug: CPX-351 (Cytarabine:Daunorubicin) Liposome Injection

SUMMARY:
The primary objective of this study is to determine the recommended dose of CPX-351 for use in a phase 2 efficacy study in patients with leukemia. Secondarily, the study will assess the safety, serious adverse effects and how the body handles CPX-351. Preliminary evidence of antitumor activity will also be determined.

DETAILED DESCRIPTION:
CPX-351 is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. The two drugs are present inside the liposome in a 5:1 molar ratio. The development of CPX-351 (cytarabine:daunorubicin) Liposome Injection was based on 1) defining a synergistic ratio of the two active moieties, cytarabine and daunorubicin, using cell-based screening assays and 2) designing a liposomal drug carrier to maintain this ratio after intravenous administration. CPX-351 was found to be more active in in vivo models of cancer than combinations of conventional cytarabine and daunorubicin. Both cytarabine and daunorubicin are active chemotherapeutic agents, each approved for clinical use in the United States for the treatment of hematological neoplasms.

CPX-351 is being developed with the hypothesis that it is superior to the currently used regimen of cytarabine and daunorubicin in the treatment of acute leukemia. This phase I study will determine the dose to carry forward into phase II trials.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Age > 18 years at the time of signing the informed consent form
* Pathological confirmation of leukemia or myelodysplastic syndrome.
* AML according to WHO criteria; except for core-binding factor AMLs (t(8;21), inv(16) or t(16;16)) and APL
* ALL
* MDS
* Patients with AML include the following:
* Patients in 2nd or greater relapse
* Patients in first relapse with initial CR duration lasting <6 months
* Patients in first relapse refractory to induction therapy
* Patients with primary refractory AML
* Patients with ALL include the following
* Patients with T-cell ALL refractory or in relapse following nelarabine
* Patients with other ALL that is refractory or in relapse.
* Patients with MDS include the following:
* The subset of RAEB-2 patients with >10% blasts with at least 1 prior therapy that includes a hypomethylating agent.
* Previously untreated chemotherapy induced AML
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0,1 or 2
* Able to adhere to the study visit schedule and other protocol requirements
* Life expectancy of at least 12 weeks
* Laboratory values fulfilling the following:
* Serum creatinine < 1.5 mg/dL
* Serum total bilirubin < 1.5 mg/dL
* Serum alanine aminotransferase or aspartate aminotransferase < 150 IU/liter Note: If elevated liver enzymes are related to disease; contact medical monitor to discuss.
* Cardiac ejection fraction > 50% by MUGA scan or echocardiography
* All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the patient from signing the informed consent form
* Chemotherapy or other investigational anticancer therapeutic drugs in the two weeks prior to study entry; in the event of rapidly proliferative disease, however, the use of hydroxyurea is permitted up to 24 hours before study entry
* Clinical evidence of active CNS leukemic involvement
* Pregnant or lactating women
* Clinically significant cardiac disease (New York Heart Association Class III or IV)
* Severe debilitating pulmonary disease
* Active and uncontrolled infection. Patients with an infection under active treatment with antibiotics and whose infection is controlled may be entered into the study
* Current evidence of invasive fungal infection (blood or tissue culture); HIV or hepatitis C infection
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-related disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) for use in phase 2

SECONDARY OUTCOMES:
To evaluate the safety and dose-limiting toxicities (DLT) of CPX-351.
To determine the pharmacokinetic parameters of CPX-351 administered in this schedule.
To assess preliminary efficacy information of CPX-351 administered in this schedule in patients with advanced leukemias.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Louie, M.D., Study Director — Jazz Pharmaceuticals; Jonathan Kolitz, M.D., Principal Investigator — New York School of Medicine at North Shore University Hospital
Locations (4):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffit Cancer Center & Research Institute at the University of S. Florida, Tampa, Florida
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital Weill Medical College of Cornell University, New York, New York

REFERENCES:
- [Derived] Feldman EJ, Kolitz JE, Trang JM, Liboiron BD, Swenson CE, Chiarella MT, Mayer LD, Louie AC, Lancet JE. Pharmacokinetics of CPX-351; a nano-scale liposomal fixed molar ratio formulation of cytarabine:daunorubicin, in patients with advanced leukemia. Leuk Res. 2012 Oct;36(10):1283-9. doi: 10.1016/j.leukres.2012.07.006. Epub 2012 Jul 26. PMID 22840315